CLINICAL TRIAL: NCT03330184
Title: Effectiveness and Safety of Berberine Hydrochloride and Bifidobacterium in People With Abnormal Glucose Level: an Multicenter, Randomized, Double-blinded, Placebo-controlled Study.
Brief Title: Effectiveness and Safety of Berberine Hydrochloride and Bifidobacterium in People With Abnormal Glucose Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Second Affiliated Hospital of Xi'an Jiaotong University (Other); Yan'an University Affiliated Hospital (Other); Shaanxi Aerospace Hospital (Unknown); Genertec Universal Xi'an Aero-Engine hospital (Xi' an) Co., Ltd (Unknown); Xi'an Gaoxin Hospital (Other); Chang'An Hospital (Other); Xi'an Central Hospital (Other); Yan'an people's Hospital (Unknown); Shangluo Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013KTZB
Record Dates: First submitted 2017-10-18; First posted 2017-11-06 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2018-11

CONDITIONS: Berberine Hydrochloride
Keywords: Bifidobacterium; People With Abnormal Glucose Level

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Berberine Hydrochloride group (Experimental): 2/day, 16 weeks
  Interventions: Drug: Berberine Hydrochloride group
- Bifidobacterium group (Experimental): 2/day, 16 weeks
  Interventions: Drug: Bifidobacterium group
- Berberine Hydrochloride and Bifidobacterium group (Experimental): 2/day, 16 weeks
  Interventions: Drug: Berberine Hydrochloride and Bifidobacterium group
- placebo (Placebo Comparator): bifidobacterium mimetic capsules berberine mimetic tablets,2/day, 16 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Berberine Hydrochloride group
  Arms: Berberine Hydrochloride group
Drug: Bifidobacterium group
  Arms: Bifidobacterium group
Drug: Berberine Hydrochloride and Bifidobacterium group
  Arms: Berberine Hydrochloride and Bifidobacterium group
Drug: placebo
  Arms: placebo

SUMMARY:
The aim of this study is to assess the beneficial effects of Bifidobacterium and Berberine Hydrochloride on lowering glucose and delaying progress to diabetes in patients with prediabetes and to detect the potential mechanism.

DETAILED DESCRIPTION:
Gut microbiota may play an important role in patients with prediabetes. Berberine, which is usually used as an antibiotic drug, has been reported a potential glucose-lowering effect in vitro and in vivo studies. Bifidobacterium, as a familiar probiotics, can modulate gut microbiota and improve glucose and lipid metabolism in animal experiments. Therefore, the aim of this study is to assess the beneficial effects of Bifidobacterium and Berberine Hydrochloride on lowering glucose and delaying progress to diabetes in patients with prediabetes and to detect the potential mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities.
* Male or female between 18 and 70 years of old.
* 19≤Body mass index(BMI)≤30kg/m^2.
* No participate in any clinical trial at least 3 months.
* Diagnosed impaired fasting glucose(IFG) and impaired glucose tolerance(IGT) or Diabetes.
* In visit 1, 5.60mmol/L≤Fasting plasma glucose(FPG)<8.0mmol/L; in visit 2, 6.1≤FPG<8.0mmol/L or 7.8≤2-hour postprandial plasma glucose(2h-PPG) <17mmol/L.
* Females in child-bearing period should be given birth control.
* No severe disease about heart, lung and kidney.

Exclusion Criteria:

* Type 1 diabetes
* Diabetes patients with previously treated or untreated FPG ≥ 8 mmol/L or 2-h PPG ≥ 17 mmol/L;
* Women of childbearing potential who are pregnant, breastfeeding or intend to become pregnant or are not using adequate contraceptive methods.
* Those who are allergic to study drugs
* Unable to cooperate
* Abnormal liver function, ALT and AST are more than 2 times of the normal upper limit
* Renal injury, blood creatinine ≥133 µmol/L
* Poor blood pressure control, systolic blood pressure SBP≥160mmHg and/or diastolic blood pressure DBP≥95mmHg
* Patients with chronic gastrointestinal diseases (pancreatitis, inflammatory bowel disease) and history of intestinal surgery
* Patients with severe heart disease, such as heart failure, unstable angina pectoris, acute myocardial infarction
* Chronic hypoxic diseases such as emphysema, pulmonary heart disease
* Having obvious diseases of the blood system
* Persons with tumor diseases
* Endocrine diseases, such as hyperthyroidism and hypercortisolism
* Mental illness, abuse of alcohol, drugs or other substances
* Persons with long-term oral or intravenous corticosteroid hormones therapy
* Having stress conditions such as surgery, severe trauma, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change of absolute value of fasting plasma glucose (mmol/L) | baseline and week 16
  Fasting plasma glucose will be measured during oral glucose tolerance test (OGTT) by glucose oxidase method at baseline and week 16.

SECONDARY OUTCOMES:
Change of absolute value of 2-hour postprandial plasma glucose (mmol/L) | baseline and week 16
  2-hour postprandial plasma glucose will be measured during OGTT by glucose oxidase method at baseline and week 16.
Change of level of HbA1c (%) | baseline and week 16
  HbA1c will be tested in plasma by high-performance liquid chromatography at baseline and week 16.
Change of level of systolic pressure (mmHg) | baseline and week 16
  Systolic pressure will be measured by mercurial sphygmomanometer using the standard methods at baseline and week 16.
Change of level of diastolic pressure (mmHg) | baseline and week 16
  Diastolic pressure will be measured by mercurial sphygmomanometer using the standard methods at baseline and week 16.
Change of level of serum total cholesterol (mmol/L) | baseline and week 16
  Serum total cholesterol will be measured by fully automatic biochemical analyser at baseline and week 16.
Change of level of low-density lipoprotein cholesterol (mmol/L) | baseline and week 16
  Serum low-density lipoprotein cholesterol will be measured by fully automatic biochemical analyser at baseline and week 16.
Change of level of high-density lipoprotein cholesterol (mmol/L) | baseline and week 16
  Serum high-density lipoprotein cholesterol will be measured by fully automatic biochemical analyser at baseline and week 16.
Change of level of triglycerides (mmol/L) | baseline and week 16
  Serum triglycerides will be measured by fully automatic biochemical analyser at baseline and week 16.
Change of absolute value of body weight (kg) | baseline and week 16
  Body weight will be measured by weighing scale using the standard methods at baseline and week 16.
Change of absolute value of body mass index (BMI) (kg/m^2) | baseline and week 16
  Weight and height will be combined to report BMI in kg/m^2 at baseline and week 16.
Change of level of homeostasis model assessment (HOMA) index | baseline and week 16
  Fasting serum insulin and fasting plasma glucose will be calculated for HOMA index at baseline and week 16.
Change of level of insulin early-phase secretion index | baseline and week 16
  Fasting serum insulin and 30 min post serum insulin during OGTT will be calculated for early-phase secretion index at baseline and week 16 .
Change of level of insulin late-phase secretion index | baseline and week 16
  Fasting serum insulin and 2-hour post serum insulin during OGTT will be calculated for late-phase secretion index at baseline and week 16 .
Change of level of GLP-1(pmol/L) | baseline and week 16
  GLP-1 will be measured in serum by ELISA KIT at baseline and week 16.
Change of abundances of gut microbiota (%) | baseline and week 16
  Fecal samples will be measured by metagenomic sequencing to obtain abundances of gut microbiota at baseline and week 16.

CONTACTS AND LOCATIONS:
Overall Officials: Qiuhe Ph.D. Ji, M.D., Principal Investigator — Department of Endocrinology,Xi jing Hospital,Fourth Military Medical University

REFERENCES:
- [Derived] Ming J, Yu X, Xu X, Wang L, Ding C, Wang Z, Xie X, Li S, Yang W, Luo S, He Q, Du Y, Tian Z, Gao X, Ma K, Fang Y, Li C, Zhao J, Wang X, Ji Q. Effectiveness and safety of Bifidobacterium and berberine in human hyperglycemia and their regulatory effect on the gut microbiota: a multi-center, double-blind, randomized, parallel-controlled study. Genome Med. 2021 Aug 9;13(1):125. doi: 10.1186/s13073-021-00942-7. PMID 34365978
- [Derived] Ming J, Xu S, Liu C, Liu X, Jia A, Ji Q. Effectiveness and safety of bifidobacteria and berberine in people with hyperglycemia: study protocol for a randomized controlled trial. Trials. 2018 Jan 26;19(1):72. doi: 10.1186/s13063-018-2438-5. PMID 29373989